CLINICAL TRIAL: NCT03245606
Title: Combining MRI Steatosis Assessment and Transient Elastography to Improve Liver Fibrosis Diagnosis in Non-Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Combining MRI Steatosis Assessment and Transient Elastography to Improve Liver Fibrosis Diagnosis in Non Alcoholic Fatty Liver Disease
Acronym: FibroMR
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_9794_FibroMR
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: NAFLD; steatosis; fibrosis; transient elastography
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Non Alcoholic Fatty Liver Disease: Patients (240) will undergo a medical examination in order to analyse their medical history and check inclusion and non-inclusion criterions.
  Then will be performed:
  * a liver biopsy
  * an abdominal MRI
  * a transient elastography
  Interventions: Procedure: Liver biopsy; Device: Abdominal MRI; Device: Transient elastography

INTERVENTIONS:
Procedure: Liver biopsy — Measurement of liver fibrosis
Device: Abdominal MRI — Measurement of liver fibrosis
Device: Transient elastography — Measurement of liver fibrosis

SUMMARY:
The main objective is to compare the accuracy of transient elastography taking into account liver steatosis determined by MRI, to liver biopsy for the diagnosis of liver fibrosis ≥F2 in patient with NAFLD.

DETAILED DESCRIPTION:
No alcoholic fatty liver disease (NAFLD) is induced by an abnormal build up of fat in the liver. It can induce liver damage, namely fibrosis, which leads to cirrhosis and an increased risk of liver cancer. The diagnosis of liver fibrosis is thus critical to identify patients at risk.

Liver biopsy is the gold standard for the diagnosis of liver fibrosis. However this invasive test is expensive and has a significant morbidity.

To avoid this others non invasive test have been developed to assess steatosis and fibrosis of the liver :

* Magnetic Resonance Imaging can quantify liver steatosis accurately.
* Transient elastography (Fibroscan®) is approved for the diagnosis of fibrosis in chronic hepatitis C. However results in NAFLD were disappointing. Further, steatosis by heightening liver elasticity is thought to be the cause of these poor results.
* Several biological tests or score are also approved in chronic hepatitis C, but not in NAFLD.

The hypothesis driving this study is that by accounting for liver steatosis through the mean of MRI, we could more accurately interpret transient elastography value to accurately diagnose the severity of liver fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* For which a liver biopsy is indicated for NAFLD according to current guidelines
* Presenting with at least one of the metabolic syndrome criteria:

  * BMI > 25 kg/m² and/or Waist circumference ≥ à 94cm for men / ≥ à 80cm for women
  * Fasting glucose > or = to 5,6 mmol/L or diabetes / or lowering glucose treatment
  * Blood pressure ≥ 130/85 mmHg / or treatment
  * Triglycerides ≥ than 1,7 mmol/L
  * HDL-C ≤ than 1 mmol/L (men), ≤ 1,3 mmol/L (women) /or lipid lowering treatment
* Affiliated to medical care insurance
* Having signed informed consent for participating in the study

Exclusion Criteria:

* Associated other chronic liver disease : infectious, auto immune, genetic
* Alcohol consumption higher than 21 standard unit per week for men, or 14 standard unit for women;
* Steatosis inducing treatment: steroids, amiodarone, methotrexate, tamoxifen
* History of bariatric surgery
* Contra indication to MRI (pace maker, metallic foreign body, claustrophobia)
* Persons subject to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NAFLD
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Comparison of the accuracy of transient elastography taking into account liver steatosis determined by MRI, to liver biopsy for the diagnosis of liver fibrosis ≥F2 in patient with NAFLD | Day 1
  Determination of the fibrosis stage by a double blind reading of liver biopsy by experienced pathologist

SECONDARY OUTCOMES:
Assessment of accuracy of transient elastography corrected according to the degree of liver steatosis determined by MRI for the diagnosis of liver fibrosis ≥F2 in patient with NAFLD compared to liver biopsy | Day 1
Assessment of accuracy of transient elastography taking into account liver steatosis determined by MRI, for the diagnosis of liver fibrosis at all fibrosis stage (F1-F2-F3-F4) in patient with NAFLD compared to liver biopsy | Day 1
Assessment of accuracy of transient elastography corrected according to the degree of liver steatosis determined by MRI for the diagnosis of liver fibrosis at all fibrosis stage (F1-F2-F3-F4) in patient with NAFLD compared to liver biopsy | Day 1
Assessment of accuracy of Acoustic Radiation Force Impulse for the diagnosis of liver fibrosis ≥F2 in patient with NAFLD compared to liver biopsy | Day 1

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHU d'Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - CHD Vendée, La Roche-sur-Yon
  - Groupe Hospitalier Bretagne Sud, Lorient
  - CHU de Nantes, Nantes
  - CHU de Rennes, Rennes
  - CH de Saint Brieuc, Saint-Brieuc
  - CHU de Toulouse, Toulouse
  - Centre Hospitalier Bretagne Atlantique, Vannes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Masrour O, Ehrhard F, Guillaume M, Boursier J, Gournay J, Aziz K, Schnee M, Garlantezec R, de Ledinghen V, Morcet J, Laine F, Allaume P, Turlin B, Gandon Y, Bardou-Jacquet E. Diagnostic accuracy of transient elastography in MASLD is independent of MRI-PDFF steatosis in a multicenter study. JHEP Rep. 2025 Sep 11;7(12):101589. doi: 10.1016/j.jhepr.2025.101589. eCollection 2025 Dec. PMID 41334457